CLINICAL TRIAL: NCT06987877
Title: Prospective Randomized Controlled Trial Evaluating the Efficacy of Routine Saline Flushing in the Prevention of Nephrostomy Tube Obstructions: A Pilot Study
Brief Title: Efficacy of Routine Saline Flushing in the Prevention of Nephrostomy Tube Obstructions: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Yan Epelboym, M.D.,M.P.H., Assistant Professor of Radiology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024p003079
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Nephrostomy
Keywords: Nephrostomy occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Flushing of Nephrostomy (Active Comparator): Subjects in the routine flushing group will continue to flush their nephrostomy tubes once per day with 10mL of normal saline
  Interventions: Other: Flushing of nephrostomy
- No Flushing of Nephrostomy (Experimental): Subjects allocated to the study intervention group will not flush their nephrostomy tube during the duration of the research study
  Interventions: Other: No flushing of the nephrostomy

INTERVENTIONS:
Other: No flushing of the nephrostomy — Subjects allocated to the study intervention group will not flush their nephrostomy tube during the duration of the research study
  Arms: No Flushing of Nephrostomy
Other: Flushing of nephrostomy — Subjects assigned to this cohort will flush their nephrostomy catheter once daily with 10 mL of normal saline
  Arms: Routine Flushing of Nephrostomy

SUMMARY:
The investigators performing this research to study if routine flushing is necessary to prevent obstructions of a nephrostomy tube. This study will evaluate patients that have nephrostomy tube or will have nephrostomy tubes placed as part of their standard clinical care.

If participants agree to participate in this study, participants will undergo randomized assignment to either continue to routinely flush the nephrostomy tube with normal saline or not to routinely flush the nephrostomy tube with normal saline. Participantswill be in the study for approximately 3 months if they decide to stay for the whole study.

DETAILED DESCRIPTION:
A percutaneous nephrostomy tube (PCN) is an external draining catheter that is positioned within the renal pelvis to allow urine to drain externally. PCNs may be placed for several indications including for urinary obstruction, urinary diversion, or to create an access point for endoscopic procedures. Patients often return to the interventional suite prior to their routine preventative exchange due to catheter related complications, such as dislodgement, kinking, or blockages. Often, these catheter related complications require additional procedures, which adds risk from instrumentation and sedation.

Routine saline flushing of percutaneous nephrostomy tubes is commonly performed at many institutions with the intent of reducing incidences of tube obstruction. Patients at some institutions are instructed to flush their nephrostomy tubes between one to three times a day with 10mL of normal saline. Although routine flushing is widely practiced, to our knowledge, there is no published evidence to support the efficacy of flushing in reducing incidence of nephrostomy tube obstruction. Furthermore, flushing of the percutaneous nephrostomy tubes may impact patient's quality of life, due to discomfort related with flushing, bear cost to the patient, and manipulation of the catheter while flushing, which may lead to inadvertent dislodgment.

In this pilot study, the investigators would like to investigate if there is any significant difference of routine flushing of nephrostomy tubes on the rates of nephrostomy tube obstructions. If there is no significant difference, this could potentially lead to larger studies that can elucidate the efficacy of this practice.

Normal Saline Normal saline is an isotonic solution of 0.9% of sodium chloride and contains 154 mmol/L of sodium and chloride ions. It widely used intravenously for fluid resuscitation or as a drug solvent. Intravenous administration of normal saline has very little impact on the human body in patients with normal renal function and in physiologic conditions. In addition, it has also been used to flush a wide variety of catheters in the interventional radiology field, including abscess drains, percutaneous biliary drains, and nephrostomy tubes. Any impact of normal saline administered directly into the urinary system has never been studied, although it has been thought to be safe and is commonly performed in interventional radiology practice.

Proposed Research

The investigators hypothesize that routine flushing of percutaneous nephrostomy tubes does not significantly change the incidence of nephrostomy tube obstructions. The study design is a single center, prospective, randomized pilot study. The investigators will enroll 20 patients with nephrostomy tubes, male, female, or non-binary, aged 18 - 80 years, with a new or ongoing indication for a nephrostomy tube. Subjects will be allocated 1:1 to the intervention, no routine flushing of the nephrostomy tube, and control arms, routine flushing of the nephrostomy tube. Any patients who are on a shortened exchange interval due to frequent encrustations of their nephrostomy tubes or have a planned definitive treatment for the indication of their nephrostomy tube prior to their next scheduled routine exchange will be excluded.

Patients will be enrolled at their index nephrostomy tube placement or their routine nephrostomy tube exchange. Once enrolled, the patients will undergo randomization to either the experimental or control arms. The patient will then undergo the percutaneous nephrostomy tube placement or exchange procedure per standard of care. There will be a single follow up timepoint at their routine exchange appointment or earlier if there are any catheter related complications and it is determined, per standard of care, that an unplanned nephrostomy tube exchange procedure is indicated. At the follow up timepoint, a physician will determine if there is any obstruction or dislodgement of the nephrostomy tube.

ELIGIBILITY:
Inclusion Criteria:

• Age 18-80, with planned nephrostomy tube exchange or new nephrostomy tube placement with ongoing need for a nephrostomy tube.

Exclusion Criteria:

* Current local infection
* History of anaphylaxis to iodinated contrast
* Pregnant or intent to become pregnant during the study
* Irreversible coagulopathy
* Planned for definitive treatment for the clinical indication of the nephrostomy tube prior to 12-week post-intervention.
* Planned routine exchange prior to 12 weeks after nephrostomy tube exchange or placement procedure
* Complete sensory loss below T10 dermatome.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Tube Obstruction | 12 weeks
  The primary endpoint is the difference in rate of nephrostomy tube obstructions prior to 12-week routine maintenance exchanges in the intervention and control groups.

SECONDARY OUTCOMES:
Tube Dislodgement | 12 weeks
  The secondary endpoint is the difference in rates of clinically significant dislodgement between the routine flushing group and the non-routine flushing groups defined as any retraction of the nephrostomy tube requiring an unscheduled nephrostomy tube exchange due to catheter malfunction prior to a routine maintenance exchange at 12-weeks post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Epelboym, MD, MPH, Principal Investigator — MGB
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Demographics Tube occlusion rates Tube dislodgement rates